CLINICAL TRIAL: NCT04592965
Title: Unravelling Dysfunctional Brain Networks in Patients With Parkinson's Disease Suffering From Hallucinations
Brief Title: Hallucinations in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olaf Blanke (Other)
Collaborators: University Hospital, Geneva (Other); Hôpital du Valais (Other); Insel Gruppe AG, University Hospital Bern (Other); Centre Hospitalier Universitaire Vaudois (Other); Hospital de Sant Pau (Other)
Responsible Party: Sponsor-Investigator, Olaf Blanke, Professor Doctor, Ecole Polytechnique Fédérale de Lausanne
Organization: Ecole Polytechnique Fédérale de Lausanne (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UH_PD
Record Dates: First submitted 2020-07-15; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease Psychosis
Keywords: Parkinson; fMRI; hallucinations; presence hallucination; sense of presence; connectivity
MeSH Terms: conditions — Hallucinations | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Clinical and neuropsychological examinations (Experimental): Participants will be assessed by means of validated and lab-tailored clinical scales, alongside with semi-structured interviews, to assess the status of the disease (PD), amongst others, such as cognitive capabilities.
  Interventions: Behavioral: Clinical and neuropsychological assessments
- Robot induced PH, through sensorimotor stimulation (Experimental): Participants will manipulate a patented robotic system designed to induce the PH and other accompanying bodily illusions. At the end, participants will report on various subjective experiences, by answering a structured questionnaire.
  Interventions: Behavioral: Induction of PH and associated bodily states
- Resting-state fMRI acquistion (Experimental): We will acquire resting-state data in the MRI scanner for all the participants. Respiration and heart beat rate data will also be acquired.
  Interventions: Other: Resting-state fMRI acquisition
- Robot induced PH, through sensorimotor stimulation (MRI) (Experimental): All healthy participants, and all patients who are deemed capable of performing the robotic manipulation task in the MRI scanner, will take part on this arm. Participants will perform a robotic manipulation task, with a patented robotic system, capable of inducing the PH and other accompanying bodily illusions in the MRI scanner. At the end participants will report on the various subjective experiences, by answering a structured questionnaire.
  Interventions: Other: Induction of PH and associated bodily states (MRI)

INTERVENTIONS:
Behavioral: Clinical and neuropsychological assessments — The assessment of disease state, clinical condition, and of cognitive and neuropsychological attributes.
  Arms: Clinical and neuropsychological examinations
Behavioral: Induction of PH and associated bodily states — Assessment of subjective sensitivity to the induction of the PH and associated bodily states, for different populations of PD patients and healthy aged-matched controls
  Arms: Robot induced PH, through sensorimotor stimulation
Other: Resting-state fMRI acquisition — Investigation of neural mechanisms at rest, that are potentially disrupted at different degrees, for the different clinical groups of PD patients, compared to the healthy aged-matched controls
  Arms: Resting-state fMRI acquistion
Other: Induction of PH and associated bodily states (MRI) — Assessment of subjective sensitivity to the induction of the PH and associated bodily states, for different populations of PD patients and healthy aged-matched controls Assessment and comparison of the neural mechanisms responsible for the induction of the PH and associated bodily illusions, in different groups of PD patients and healthy aged-matched controls
  Arms: Robot induced PH, through sensorimotor stimulation (MRI)

SUMMARY:
Investigation on how robotically mediated sensorimotor stimulation induces and triggers presence hallucinations in different clinical groups of parkinsonian patients, and in aged-matched controls

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a condition mostly known and characterized by motor symptoms, such as tremors, rigidity, bradykinesia, amongst others. Yet, recent bodies of research have identified a significant number of non-motor symptoms that also accompany the unfolding of this disease. These non-motor symptoms mainly focus on hallucinations that will develop with the course of the disease, and will affect approximately 50% of the patients suffering from Parkinson's. This number rises to 70% if minor hallucinations, mild phenomena and poorly-structured hallucinations, are included. Despite the potential impact in the patients' lives, and previous efforts to study these phenomena, the brain changes that underly hallucinations in PD are still poorly understood. With the current study the investigators aim to improve this understanding, by studying the most common minor hallucination in Parkinson's Disease, the Presence Hallucination (PH), which can be defined as the strange sensation of perceiving someone behind when no one is actually there. To study it in a controlled manner, the investigators will induce this hallucination with an extensively verified paradigm, which gives rise to this sensation through robotically-mediated sensorimotor stimulation, in both healthy individuals, and PD patients. The researchers intend to discern the sensitivity of different groups of PD patients to the induction of this hallucination, by targeting PD patients, with hallucinations including PH, with hallucinations but without PH, without any hallucinations, and an aged match control group with no neurological comorbidities. The investigators intended to extend previous work on the induction of the PH in PD patients, by identifying the neural correlates of this induction in these patients, in a similar fashion to previous work in healthy individuals. Moreover, the researchers also intend to extend the general understanding of the basis for hallucinations in PD by extending what was done in previous work, to more stratified cohorts of PD patients, that will not only be analysed in terms of static during rest, but also in terms of dynamic connectivity, and will also perform the PH-inducing task in the scanner, as mentioned before.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease (expect for healthy controls)
* Able to understand instructions and provide informed consent.
* Native speaking language of experimental site (or acquisition of language of experimental site before 6 years old).
* Montreal Cognitive Assessment (Nasreddine & Patel, 2016) with score ≥ 22.
* Able to manipulate the robotic device.

Exclusion Criteria:

* For PD patients only: Neurological comorbidities other than Parkinson's disease (e.g. Alzheimer's disease, vascular dementia, multiple sclerosis, stroke, traumatic brain injury, epilepsy, chronic migraine, etc.)
* For healthy controls only: Parkinson's disease or other neurological illnesses
* History or current condition of substance abuse and/or dependence (e.g., alcohol, drugs).
* Suffering from or diagnosed with psychiatric illnesses according to DSM-V criteria (e.g., schizophrenia, bipolar disorders, autism, personality disorders, phobia etc.).
* Family history (1st and 2nd degree) of psychiatric disorders (e.g., schizophrenia or bipolar disorders).
* Severe somatic illnesses (e.g., cancer).
* Severe tremors or physical disability preventing optimal use of robotic device.
* Participating in a pharmacological study.
* Local or general anaesthesia 30 days prior experiment
* Inability to provide informed consent (legal guardianship)
* For the MRI part only: body weight exceeding 160kg, implanted metallic devices, implant for deep brain stimulation, foreign metallic objects, unstable angina, cardio-vascular diseases, tattoos with metallic components, external metallic objects, claustrophobia, pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity to the induction bodily illusions of Presence Hallucination, Passivity experiences, loss of agency, and control questions, through lab-tailored questionnaires (7-point Likert-scale) | 5 minutes, at the end of each participant's session in arm 2
  Note that for the measuring the sensitivity of each patient to the induction of the presence hallucination, passivity sensations, loss of agency, and control questions, the patients will perform two manipulations with the robotic system described in the introduction, in both the synchronous and asynchronous conditions
Sensitivity to the induction bodily illusions of Presence Hallucination, Passivity experiences, loss of agency, and control questions, through lab-tailored questionnaires (7-point Likert-scale) in the MRI scanner | 5 minutes, at the end of each participant's session in arm 4
  After the sensorimotor task in the MRI scanner that induces the presence hallucination, ratings for the strength of the perceived sense of presence and associated phenomena are collected with the participants
fMRI blood-oxygen level dependent signal response during resting state | Approximately 30 minutes, during arm 3
  We will analyse resting state data from the different populations of PD patients in this study and healthy controls
fMRI blood-oxygen level dependent signal during robotic stimulation | Approximately 45 minutes, during arm 4
  We will analyse neural data from PH-induction inside the scanner, from the different populations of PD patients in this study and healthy controls

SECONDARY OUTCOMES:
Dosage of dopaminergic medication (in daily equivalent mg/day) | Approximately 10 minutes during screening
  Dosage of dopaminergic medication (in daily equivalent mg/day)
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 15 minutes during arm 1
  The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale provides assessment of both motor and non-motor symptoms experienced by the patients during the last 7 days prior the examination. The scale comprise both self-report and semi-structured evaluations. The severity of each symptom is measured on a Likert-type scale from 0 (normal) to 4 (severe). Therefore the higher the score, the more impaired is the patient. The MDS-UPDRS has 50 items, categorised into four parts, namely, I: Non-motor experiences of daily living (range 0-52) II: Motor experiences of daily living (range 0-52) III: Motor examination (range 0-124) IV: Motor complications (range 0-24) I: Non-motor experiences of daily living II: Motor experiences of daily living III: Motor examination IV: Motor complications
Scale for the Assessment of Positive Symptoms (SAPS) | 15 minutes during arm 1
  The SAPS is a validated clinical rating scale measuring positive symptoms of schizophrenia, recommended by the MDS to assess psychotic symptoms in PD, in the absence of a reliable validated one. The scale is sub-categorised into 4 domains within which specific symptoms are evaluated from 0 (absent) to 5 (severe): Hallucinations (67 items + 1 global evaluation item) (e.g., visual, auditory) (range 0-30); Delusions (12 items + 1 global evaluation item) (e.g., persecution, thought insertion) (range 0-60); Bizarre behaviour (4 items + 1 global evaluation item) (e.g., agitation, social behaviour) (range 0-20); Positive formal thought disorder (8 items+ 1 global evaluation item) (e.g., incoherence) (range 0-40) A composite score is calculated by adding the scores of each non-global item.. A global score of severity of symptoms with regard to duration and persistence of symptoms can be calculated by adding the scores of the global evaluation items.
Hallucination questionnaire specific for PD | 15 minutes during arm 1
  This questionnaire is based on previous lab research and is a semi-structured interview on hallucinations and other psychotic symptoms. The frequency of symptoms is evaluated on a scale from 0 to 4. Two scoring systems are proposed to evaluate severity of symptoms (from 1-3): Severity score 1 refers to the impact of the symptoms on the patients' environment (ex: caregivers, family) as defined by the patients; Severity score 2 refers to the clinical severity as estimated by the clinician during the clinical interview. A composite score for each symptom is calculated: Frequency x Severity 1 (and Frequency x Severity 2). The composite scores of each symptom are then added to obtain the total score for the Category. The total score of the full scale is calculated by adding the total scores of Category A to E. The greater the score, the more frequent and severe the symptoms are.
The Hospital Anxiety and Depression Scale (HADS) | 5 minutes during arm 1
  The Hospital Anxiety and Depression Scale is a 14-item self-assessment scale found to be a reliable instrument for detecting states of depression and anxiety. Seven items are dedicated to assess anxiety and the 7 others for depression on a 4-point Likert scale from 0 to 3.. A score > greater than 11/21 for each domain (anxiety or depression) indicates a considerable symptomatology for depression or anxiety.
REM Sleep Behaviour Disorder Screening Questionnaire (RBDSQ) | 5 minutes during arm 1
  The REM Sleep Behaviour Disorder Screening Questionnaire is a self-report 13-item questionnaire assessing clinical features of REM sleep, and is a potential marker for PD. A "yes" (score 1) or "no" (score 0) is provided for each item. A maximum score of 13 indicates severe REM sleep behaviour disorders.
Beck Cognitive Insight Scale (BCIS) | 3 minutes during arm 1
  a 15-item self-report questionnaire assessing the cognitive processes involved in the re-evaluation of anomalous experiences and their misinterpretations, i.e., distancing, objectivity, perspective, and self-correction. Subjects will rate on a scale from 0 (do not agree at all) to 3 (agree completely) how much they agree with each statement. A general insight ratio can also be calculated: self-reflectiveness sore/self-certainty score. High score reflects better cognitive insight (max=6).
UCLA loneliness questionnaire | 2 minutes during arm 1
  This is a 3-item scale assessing the overall subjective feeling of loneliness in elderly populations from 1 (hardly) to 3 (often). A maximum score of 9 indicates the highest level of subjective feeling of loneliness.
Dimensional Apathy Scale (DAS) | 5 minutes during arm 1
  The Dimensional Apathy Scale is a 24-item self-report questionnaire assessing three apathetic subtypes; namely cognitive, emotional-affective and auto-activation apathy. Subjects rate on a scale from 0 (almost always) to 3 (hardly ever) how much they agree with each statement. The scale provides the following sub-scores: (1) executive subscale, (2) emotional subscale and (3) behaviour/cognitive initiation subscale. A total score can be calculated. The maximum of each sub-scale is 24 and the total is 72. The cut-off score for each sub-scale are as follows:
  Executive: 14 Emotional: 15 Initiation: 16 Scoring below the cut-off indicates substantial clear apathetic symptoms.
Questionnaire for Impulsive-compulsive Disorders in Parkinson's Disease (QUIP) | 5 minutes during arm 1
  The Questionnaire for Impulsive-compulsive Disorders in Parkinson's Disease self-rating assesses 7 major behaviours :1. Gambling, 2. Sex, 3. Buying, 4. Binge eating, 5. Hobbyism, 6. Punding and 7. Excessive medication use. Each behaviour is assessed by means of 4 questions on a Liket type scale from 0 (never) to 4 (very often). The scores of for each behaviour range from 0-16, and the total score to the scale ranges from 0-112. High scores reveal impulsive-compulsive disorders.
Neuropsychiatric Fluctuations Scale for Parkinson's Disease (NPS) | 5 minutes during arm 1
  The Neuropsychiatric Fluctuations Scale for Parkinson's Disease is a 20-item self-report questionnaire. Ten items represent neuropsychiatric symptoms typically reported by patients in the OFF-medication condition and ten items measure neuropsychological symptoms typically reported by patients in the ON-medication condition. Subjects rate on a scale from 0 (no) to 3 (a lot) how much they agree with each statement. The scale provides two sub-scores, one for the ON-Items and one for the OFF-Items, ranging from 0-30. High scores indicate either ON-behaviours corresponding to ON-states (eg. euphoria, excitement) or OFF-states behaviours such as anxiety, lack of energy and fatigue.
Parkinson's disease - Cognitive Rating Scale (PD-CRS) | 25 minutes during arm 1
  Parkinson's disease - Cognitive Rating Scale is a battery of neuropsychological tests specifically designed to capture the whole spectrum of cognitive impairment in patients with PD. This battery provides, as stated by the Movement Disorders Society:
  * Frontal subcortical tasks (sustained attention, working memory, alternating and action verbal fluency, clock drawing, immediate and delayed free recall verbal memory). Scores range from 0-104.
  * Posterior cortical tasks (confrontation naming and clock copying), with scores ranging from 0 to 30.
  * Total scores range from 0-134 High scores are indicative of preserved cognitive functions.
Semantic and phonemic verbal fluency | 4 minutes during arm 1
  Within 2 minutes, participants generate orally as many animal names as possible for the semantic fluency task, and as many words starting with letter P for the phonemic task, while respecting the following rules: no repetition and no word with the same root, and no proper nouns. The total number of words correctly named, and the number of errors are taken into account. Z-scores will be calculated.
Modified 5-point test (non-verbal fluency) | 3 minutes during arm 1
  The test consists of squares containing 5 dots (like the number five on a dice). Participants are instructed to draw as many different patterns as possible, within 3 minutes, by connecting the dots by means of straight lines. The number of unique designs (maximum=80) and errors are counted. Z-scores will be calculated.
Trail Making Test A and B (TMT A; TMT B) | maximum of 3 minutes during arm 1
  The Trail Making Test is a test during which the execution of the task is timed. The time taken to complete the test are noted as well as the number of errors. Z-scores will be calculated.Part A explores perceptual-motor speed (visuo-motor tracking) while part B requires more psychomotor speed and working memory.
Symbol search | 2 minutes during arm 1
  This sub-test, derived from the Wechsler Adult Intelligence Scale, assesses visuo-motor information processing speed within 2 minutes. Participants scan a search group and indicate whether one of the non-verbal symbols in the target group matches. The raw scores obtained are converted to standard scores with respect to participant's age. Cuff off of standard score = 10. Scores below 10 are considered under the normal range.

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Blanke, Principal Investigator — Ecole Polytechnique Fédérale de Lausanne
Locations (6):
- Hospital de la Santa Creu I Sant Pau, Barcelona, Spain
- Switzerland (5):
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Inselspital, Bern
  - Campus Biotech, Geneva
  - Geneva University Hospital, Geneva
  - Hôpital du Valais, Sion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalia LV, Lang AE. Parkinson's disease. Lancet. 2015 Aug 29;386(9996):896-912. doi: 10.1016/S0140-6736(14)61393-3. Epub 2015 Apr 19. PMID 25904081
- [Background] Postuma RB, Berg D. Advances in markers of prodromal Parkinson disease. Nat Rev Neurol. 2016 Oct 27;12(11):622-634. doi: 10.1038/nrneurol.2016.152. PMID 27786242
- [Background] Wood RA, Hopkins SA, Moodley KK, Chan D. Fifty Percent Prevalence of Extracampine Hallucinations in Parkinson's Disease Patients. Front Neurol. 2015 Dec 21;6:263. doi: 10.3389/fneur.2015.00263. eCollection 2015. PMID 26733937
- [Background] Ffytche DH, Aarsland D. Psychosis in Parkinson's Disease. Int Rev Neurobiol. 2017;133:585-622. doi: 10.1016/bs.irn.2017.04.005. Epub 2017 Jun 16. PMID 28802934
- [Background] Diederich NJ, Fenelon G, Stebbins G, Goetz CG. Hallucinations in Parkinson disease. Nat Rev Neurol. 2009 Jun;5(6):331-42. doi: 10.1038/nrneurol.2009.62. PMID 19498436
- [Background] Lenka A, Pagonabarraga J, Pal PK, Bejr-Kasem H, Kulisevsky J. Minor hallucinations in Parkinson disease: A subtle symptom with major clinical implications. Neurology. 2019 Aug 6;93(6):259-266. doi: 10.1212/WNL.0000000000007913. Epub 2019 Jul 9. PMID 31289146
- [Background] Fenelon G, Soulas T, Cleret de Langavant L, Trinkler I, Bachoud-Levi AC. Feeling of presence in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2011 Nov;82(11):1219-24. doi: 10.1136/jnnp.2010.234799. Epub 2011 May 7. PMID 21551471
- [Background] Blanke O, Pozeg P, Hara M, Heydrich L, Serino A, Yamamoto A, Higuchi T, Salomon R, Seeck M, Landis T, Arzy S, Herbelin B, Bleuler H, Rognini G. Neurological and robot-controlled induction of an apparition. Curr Biol. 2014 Nov 17;24(22):2681-6. doi: 10.1016/j.cub.2014.09.049. Epub 2014 Nov 6. PMID 25447995
- [Background] Pagonabarraga J, Soriano-Mas C, Llebaria G, Lopez-Sola M, Pujol J, Kulisevsky J. Neural correlates of minor hallucinations in non-demented patients with Parkinson's disease. Parkinsonism Relat Disord. 2014 Mar;20(3):290-6. doi: 10.1016/j.parkreldis.2013.11.017. Epub 2013 Dec 10. PMID 24373690
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Andreasen NC, Arndt S, Miller D, Flaum M, Nopoulos P. Correlational studies of the Scale for the Assessment of Negative Symptoms and the Scale for the Assessment of Positive Symptoms: an overview and update. Psychopathology. 1995;28(1):7-17. doi: 10.1159/000284894. PMID 7871123
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Stiasny-Kolster K, Mayer G, Schafer S, Moller JC, Heinzel-Gutenbrunner M, Oertel WH. The REM sleep behavior disorder screening questionnaire--a new diagnostic instrument. Mov Disord. 2007 Dec;22(16):2386-93. doi: 10.1002/mds.21740. PMID 17894337
- [Background] Beck AT, Baruch E, Balter JM, Steer RA, Warman DM. A new instrument for measuring insight: the Beck Cognitive Insight Scale. Schizophr Res. 2004 Jun 1;68(2-3):319-29. doi: 10.1016/S0920-9964(03)00189-0. PMID 15099613
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Radakovic R, Abrahams S. Developing a new apathy measurement scale: Dimensional Apathy Scale. Psychiatry Res. 2014 Nov 30;219(3):658-63. doi: 10.1016/j.psychres.2014.06.010. Epub 2014 Jun 19. PMID 24972546
- [Background] Weintraub D, Hoops S, Shea JA, Lyons KE, Pahwa R, Driver-Dunckley ED, Adler CH, Potenza MN, Miyasaki J, Siderowf AD, Duda JE, Hurtig HI, Colcher A, Horn SS, Stern MB, Voon V. Validation of the questionnaire for impulsive-compulsive disorders in Parkinson's disease. Mov Disord. 2009 Jul 30;24(10):1461-7. doi: 10.1002/mds.22571. PMID 19452562
- [Background] Schmitt E, Krack P, Castrioto A, Klinger H, Bichon A, Lhommee E, Pelissier P, Fraix V, Thobois S, Moro E, Martinez-Martin P. The Neuropsychiatric Fluctuations Scale for Parkinson's Disease: A Pilot Study. Mov Disord Clin Pract. 2018 Mar 23;5(3):265-272. doi: 10.1002/mdc3.12607. eCollection 2018 May-Jun. PMID 30363450
- [Background] Pagonabarraga J, Kulisevsky J, Llebaria G, Garcia-Sanchez C, Pascual-Sedano B, Gironell A. Parkinson's disease-cognitive rating scale: a new cognitive scale specific for Parkinson's disease. Mov Disord. 2008 May 15;23(7):998-1005. doi: 10.1002/mds.22007. PMID 18381647
- [Background] Ruff RM, Allen CC, Farrow CE, Niemann H, Wylie T. Figural fluency: differential impairment in patients with left versus right frontal lobe lesions. Arch Clin Neuropsychol. 1994 Jan;9(1):41-55. PMID 14589511
- [Background] Reitan RM, Hom J, Wolfson D. Verbal processing by the brain. J Clin Exp Neuropsychol. 1988 Aug;10(4):400-8. doi: 10.1080/01688638808408248. PMID 3403703
- [Background] Wechsler, D. (2008). Wechsler Adult Intelligence Scale (4th ed.). San Antonio, TX: Pearson Assessment
- [Background] Cardebat D, Demonet JF, Viallard G, Faure S, Puel M, Celsis P. Brain functional profiles in formal and semantic fluency tasks: a SPECT study in normals. Brain Lang. 1996 Feb;52(2):305-13. doi: 10.1006/brln.1996.0013. PMID 8811961
- See also: Bernasconi F, Blondiaux E, Potheegadoo J, Stripeikyte G, ..., Blanke O. (2020) Sensorimotor hallucinations in Parkinson's Disease — https://www.biorxiv.org/content/10.1101/2020.05.11.054619v1.abstract